CLINICAL TRIAL: NCT03259113
Title: EvaLuation Using Cardiac Insertable Devices And TelephonE in Hypertrophic CardioMyopathy
Brief Title: Insertable Cardiac Monitors in Hypertrophic Cardiomyopathy
Acronym: ElucidateHcm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Gävleborg (Other)
Collaborators: Abbott Medical Devices (Industry); Norrlands University Hospital (Other)
Responsible Party: Principal Investigator, Peter Magnusson, MD, Region Gävleborg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20171331
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: insertable cardiac monitor; atrial fibrillation; non-sustained ventricular tachycardia
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Consecutive insertable cardiac monitors in 30 patients with hypertrophic cardiomyopathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insertable cardiac monitor (Other): All patients will undergo monitoring using an insertable cardiac monitor (single arm)
  Interventions: Device: Insertable cardiac monitor

INTERVENTIONS:
Device: Insertable cardiac monitor — Insertable cardiac monitor (SJM Confirm Rx) subcutaneously.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is associated with sudden cardiac death and an increased risk of atrial fibrillation and subsequent embolic event. An insertable cardiac monitor will provide data on cardiac rhythm over a period of 18 months. This will provide an extended monitoring far longer than 24-48 hours of Holter monitoring as is currently usual care. Therefore, detection of arrhythmias could be used in risk stratification and decision-making with regard to offer an implantable defibrillator and anticoagulants.

DETAILED DESCRIPTION:
Detection of non-sustained ventricular tachycardia (NSVT) and atrial fibrillation (AF) using an insertable cardiac device monitor (SJM Confirm XT) which is connected to the patients smart phone and monitored for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* hypertrophic cardiomyopathy

Exclusion Criteria:

* aortic stenosis (moderate, severe)
* hypertrophic cardiomyopathy associated with metabolic disease (e.g. Fabry) and syndromes (e.g. Noonan)
* systolic heart failure
* cardiac device (previous pacemaker, implantable defibrillator )
* history of myocardial infarction
* percutaneous coronary intervention and/or coronary artery by-pass grafting
* pulmonary vein isolation, Maze surgery, ventricular tachycardia ablation, ectopic atrial tachycardia ablation
* renal clearance below 40
* malignancy or other comorbidity with less than five years life expectancy
* pregnancy of planned within 18 months
* drug addiction, severe mental disease
* not able to participate in 18 months follow-up
* 5 years risk more than 6% according HCM risk calculator of European Society of Cardiology guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-02-16 (Estimated); Study Completion 2019-04-16 (Estimated)

PRIMARY OUTCOMES:
NSVT | 18 months
  Incidence of non-sustained ventricular tachycardia (NSVT)

SECONDARY OUTCOMES:
AF | 18 months
  Incidence of atrial fibrillation (AF)

CONTACTS AND LOCATIONS:
Overall Officials: Stellan Mörner, MD PhD, Principal Investigator — Norrlands Universitetssjukhus; Peter Magnusson, MD, Principal Investigator — Region Gävleborg
Locations (1):
- Region Gavleborg, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott PM, Gimeno JR, Thaman R, Shah J, Ward D, Dickie S, Tome Esteban MT, McKenna WJ. Historical trends in reported survival rates in patients with hypertrophic cardiomyopathy. Heart. 2006 Jun;92(6):785-91. doi: 10.1136/hrt.2005.068577. Epub 2005 Oct 10. PMID 16216855
- [Background] Maron BJ, Casey SA, Hauser RG, Aeppli DM. Clinical course of hypertrophic cardiomyopathy with survival to advanced age. J Am Coll Cardiol. 2003 Sep 3;42(5):882-8. doi: 10.1016/s0735-1097(03)00855-6. PMID 12957437
- [Background] Maron BJ, Olivotto I, Spirito P, Casey SA, Bellone P, Gohman TE, Graham KJ, Burton DA, Cecchi F. Epidemiology of hypertrophic cardiomyopathy-related death: revisited in a large non-referral-based patient population. Circulation. 2000 Aug 22;102(8):858-64. doi: 10.1161/01.cir.102.8.858. PMID 10952953
- [Background] Kofflard MJ, Ten Cate FJ, van der Lee C, van Domburg RT. Hypertrophic cardiomyopathy in a large community-based population: clinical outcome and identification of risk factors for sudden cardiac death and clinical deterioration. J Am Coll Cardiol. 2003 Mar 19;41(6):987-93. doi: 10.1016/s0735-1097(02)03004-8. PMID 12651046
- [Background] Elliott PM, Sharma S, Varnava A, Poloniecki J, Rowland E, McKenna WJ. Survival after cardiac arrest or sustained ventricular tachycardia in patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 1999 May;33(6):1596-601. doi: 10.1016/s0735-1097(99)00056-x. PMID 10334430
- [Background] American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Failure Society of America; Heart Rhythm Society; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1303-38. doi: 10.1016/j.jtcvs.2011.10.019. No abstract available. PMID 22093712
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Derived] Magnusson P, Morner S. EvaLuation Using Cardiac Insertable Devices And TelephonE in Hypertrophic Cardiomyopathy (ELUCIDATE HCM): A prospective observational study on incidence of arrhythmias. J Cardiovasc Electrophysiol. 2021 Jan;32(1):129-135. doi: 10.1111/jce.14792. Epub 2020 Nov 4. PMID 33108031